CLINICAL TRIAL: NCT02830464
Title: New Biomarkers in Heart- and Renal Failure: Cohort Study for Assessing Prognosis in Acute Coronary Syndrome and Acute/Chronic Cardiovascular and Renal Failure by Means of Fibroblast Growth Factor 23
Brief Title: New Biomarkers in Heart- and Renal Failure
Acronym: IM19 Register
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: 15-151
Record Dates: First submitted 2016-07-08; First posted 2016-07-12 (Estimated); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Heart Failure; Kidney Failure
MeSH Terms: conditions — Heart Failure; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study, prognostically relevant biomarkers for cardiovascular / renal insufficiencies will be clinically evaluated, to improve the course of assessment of such disease and to gain new insights into the typical course of congestive heart failure. This is a prerequisite to allow patients to appropriate treatment as soon as possible.

DETAILED DESCRIPTION:
In recent years advances in diagnosis/ therapy in patients with acute coronary syndromes heart failure / and renal insufficiency patients could be made. However, these diseases still associated with an increased mortality rate. The diseases affecting at the same time as the heart and the kidney contribute to the deterioration in the course of the disease. An acute or chronic functional impairment of an organ, e.g. the heart, is connected to another functional impairment, such as the kidneys. In the past, different scores to the risk and prognosis assessment have been introduced measuring many different diagnostic parameters such as E.g. age, pre-existing conditions, kidney function, heart function, and laboratory values. The scores can be used for risk assessment and treatment.

For determining the prognosis of heart and kidney-failure patients, biomarkers are analyzed. Biomarkers in the blood or urine which can provide early information on a specific course of disease are called prognostic biomarkers. In this study, prognostically relevant biomarkers for cardiovascular / renal insufficiencies will be clinically evaluated, to improve the course of assessment of such disease and to gain new insights into the typical course of congestive heart failure. This is a prerequisite to allow patients to appropriate treatment as soon as possible. An important role in heart and vascular disease can be awarded the Fibroblast growth factor 23 (FGF) 23. The height of FGF23 in the blood plasma is linked with the risk of cardiovascular events occur and the beginning of dialysis patients. FGF23 goes hand in hand with the development of heart failure or with a hospitalization as a result of heart failure.

The clinical utility of biomarkers will be examined in relation to established risk scores calculated from clinical parameters, to determine whether this biomarker of bone-heart-kidney axis can extend the forecast evaluation of patients.

ELIGIBILITY:
Inclusion Criteria:

1. at least 18 years old
2. signed informed consent
3. persons who are legally competent and mentally able to follow the instructions of study personnel
4. Patient with:

   * NSTEMI myocardial infarction = non ST-segment elevation: unstable Angina pectoris (AP) / heart attack with rise of Troponin I or T, but without ST track elevation
   * STEMI = ST-segment-elevation myocardial infarction: cardiac troponin T/where to sleep and enzyme changes and attack typical ECG changes (initial ST Elevation)
   * Acute heart failure with need of hospitalisation
   * Chronic heart failure decompensation and need to the hospitalisation and need for establishing primary > 12 hours on the station IM19 (conservative intermediate care station)

Exclusion Criteria:

1. less than 18 years old
2. pregnant women and breastfeeding women
3. previous recording on an intensive care unit or transfer to an intensive care unit within 12 h after admission the IM19 station
4. death within 12 h after admission
5. persons who are housed on official or judicial order in an institution
6. persons who are in a dependency or employment relationship to the sponsor or investigator
7. chronic dialysis patients
8. persons , who at the same time take part in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Included are patients with cardiac diseases and acute hospital admission:
  * NSTEMI myocardial infarction = non ST-segment elevation: unstable AP / heart attack with rise of Troponin I or T, but without ST track elevation
  * STEMI = ST-segment-elevation myocardial infarction: cardiac troponin T/where to sleep and enzyme changes and attack typical ECG changes (initial ST Elevation)
  * Acute heart failure with need of hospitalisation
  * Chronic heart failure decompensation and need to the hospitalisation and need for establishing primary > 12 hours on the station IM19 (conservative intermediate care station)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Survival after recording on the intermediate care station | 35 days

SECONDARY OUTCOMES:
Survival after recording on the intermediate care station | 12 months
Major adverse cardiac events | 12 months
Rehospitalisation due to cardiovascular cause | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Schuh, Priv.-Doz. Dr.med., Principal Investigator — University Hospital, Aachen
Locations (1):
- University Hospital RWTH Aachen, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roger VL, Weston SA, Redfield MM, Hellermann-Homan JP, Killian J, Yawn BP, Jacobsen SJ. Trends in heart failure incidence and survival in a community-based population. JAMA. 2004 Jul 21;292(3):344-50. doi: 10.1001/jama.292.3.344. PMID 15265849
- [Background] Braunwald E. Biomarkers in heart failure. N Engl J Med. 2008 May 15;358(20):2148-59. doi: 10.1056/NEJMra0800239. No abstract available. PMID 18480207
- [Background] Tang WH, Francis GS, Morrow DA, Newby LK, Cannon CP, Jesse RL, Storrow AB, Christenson RH, Apple FS, Ravkilde J, Wu AH; National Academy of Clinical Biochemistry Laboratory Medicine. National Academy of Clinical Biochemistry Laboratory Medicine practice guidelines: Clinical utilization of cardiac biomarker testing in heart failure. Circulation. 2007 Jul 31;116(5):e99-109. doi: 10.1161/CIRCULATIONAHA.107.185267. Epub 2007 Jul 14. No abstract available. PMID 17630410
- [Background] Anwaruddin S, Lloyd-Jones DM, Baggish A, Chen A, Krauser D, Tung R, Chae C, Januzzi JL Jr. Renal function, congestive heart failure, and amino-terminal pro-brain natriuretic peptide measurement: results from the ProBNP Investigation of Dyspnea in the Emergency Department (PRIDE) Study. J Am Coll Cardiol. 2006 Jan 3;47(1):91-7. doi: 10.1016/j.jacc.2005.08.051. Epub 2005 Dec 9. PMID 16386670
- [Background] Go AS, Chertow GM, Fan D, McCulloch CE, Hsu CY. Chronic kidney disease and the risks of death, cardiovascular events, and hospitalization. N Engl J Med. 2004 Sep 23;351(13):1296-305. doi: 10.1056/NEJMoa041031. PMID 15385656
- [Background] Olauson H, Vervloet MG, Cozzolino M, Massy ZA, Urena Torres P, Larsson TE. New insights into the FGF23-Klotho axis. Semin Nephrol. 2014 Nov;34(6):586-97. doi: 10.1016/j.semnephrol.2014.09.005. PMID 25498378
- [Background] Scialla JJ, Wolf M. Roles of phosphate and fibroblast growth factor 23 in cardiovascular disease. Nat Rev Nephrol. 2014 May;10(5):268-78. doi: 10.1038/nrneph.2014.49. Epub 2014 Apr 1. PMID 24686452
- [Background] Lutsey PL, Alonso A, Selvin E, Pankow JS, Michos ED, Agarwal SK, Loehr LR, Eckfeldt JH, Coresh J. Fibroblast growth factor-23 and incident coronary heart disease, heart failure, and cardiovascular mortality: the Atherosclerosis Risk in Communities study. J Am Heart Assoc. 2014 Jun 10;3(3):e000936. doi: 10.1161/JAHA.114.000936. PMID 24922628
- [Background] Koller L, Kleber ME, Brandenburg VM, Goliasch G, Richter B, Sulzgruber P, Scharnagl H, Silbernagel G, Grammer TB, Delgado G, Tomaschitz A, Pilz S, Berger R, Mortl D, Hulsmann M, Pacher R, Marz W, Niessner A. Fibroblast Growth Factor 23 Is an Independent and Specific Predictor of Mortality in Patients With Heart Failure and Reduced Ejection Fraction. Circ Heart Fail. 2015 Nov;8(6):1059-67. doi: 10.1161/CIRCHEARTFAILURE.115.002341. Epub 2015 Aug 13. PMID 26273098
- [Background] Brandenburg VM, Kleber ME, Vervloet MG, Tomaschitz A, Pilz S, Stojakovic T, Delgado G, Grammer TB, Marx N, Marz W, Scharnagl H. Fibroblast growth factor 23 (FGF23) and mortality: the Ludwigshafen Risk and Cardiovascular Health Study. Atherosclerosis. 2014 Nov;237(1):53-9. doi: 10.1016/j.atherosclerosis.2014.08.037. Epub 2014 Aug 28. PMID 25200615
- [Background] Hu MC, Shiizaki K, Kuro-o M, Moe OW. Fibroblast growth factor 23 and Klotho: physiology and pathophysiology of an endocrine network of mineral metabolism. Annu Rev Physiol. 2013;75:503-33. doi: 10.1146/annurev-physiol-030212-183727. PMID 23398153
- [Background] Sitara D, Kim S, Razzaque MS, Bergwitz C, Taguchi T, Schuler C, Erben RG, Lanske B. Genetic evidence of serum phosphate-independent functions of FGF-23 on bone. PLoS Genet. 2008 Aug 8;4(8):e1000154. doi: 10.1371/journal.pgen.1000154. PMID 18688277
- [Background] Kestenbaum B, Sachs MC, Hoofnagle AN, Siscovick DS, Ix JH, Robinson-Cohen C, Lima JA, Polak JF, Blondon M, Ruzinski J, Rock D, de Boer IH. Fibroblast growth factor-23 and cardiovascular disease in the general population: the Multi-Ethnic Study of Atherosclerosis. Circ Heart Fail. 2014 May;7(3):409-17. doi: 10.1161/CIRCHEARTFAILURE.113.000952. Epub 2014 Mar 25. PMID 24668259
- [Background] Ix JH, Katz R, Kestenbaum BR, de Boer IH, Chonchol M, Mukamal KJ, Rifkin D, Siscovick DS, Sarnak MJ, Shlipak MG. Fibroblast growth factor-23 and death, heart failure, and cardiovascular events in community-living individuals: CHS (Cardiovascular Health Study). J Am Coll Cardiol. 2012 Jul 17;60(3):200-7. doi: 10.1016/j.jacc.2012.03.040. Epub 2012 Jun 13. PMID 22703926
- [Background] Scialla JJ, Xie H, Rahman M, Anderson AH, Isakova T, Ojo A, Zhang X, Nessel L, Hamano T, Grunwald JE, Raj DS, Yang W, He J, Lash JP, Go AS, Kusek JW, Feldman H, Wolf M; Chronic Renal Insufficiency Cohort (CRIC) Study Investigators. Fibroblast growth factor-23 and cardiovascular events in CKD. J Am Soc Nephrol. 2014 Feb;25(2):349-60. doi: 10.1681/ASN.2013050465. Epub 2013 Oct 24. PMID 24158986
- [Background] Faul C, Amaral AP, Oskouei B, Hu MC, Sloan A, Isakova T, Gutierrez OM, Aguillon-Prada R, Lincoln J, Hare JM, Mundel P, Morales A, Scialla J, Fischer M, Soliman EZ, Chen J, Go AS, Rosas SE, Nessel L, Townsend RR, Feldman HI, St John Sutton M, Ojo A, Gadegbeku C, Di Marco GS, Reuter S, Kentrup D, Tiemann K, Brand M, Hill JA, Moe OW, Kuro-O M, Kusek JW, Keane MG, Wolf M. FGF23 induces left ventricular hypertrophy. J Clin Invest. 2011 Nov;121(11):4393-408. doi: 10.1172/JCI46122. Epub 2011 Oct 10. PMID 21985788
- [Background] Gutierrez OM, Januzzi JL, Isakova T, Laliberte K, Smith K, Collerone G, Sarwar A, Hoffmann U, Coglianese E, Christenson R, Wang TJ, deFilippi C, Wolf M. Fibroblast growth factor 23 and left ventricular hypertrophy in chronic kidney disease. Circulation. 2009 May 19;119(19):2545-52. doi: 10.1161/CIRCULATIONAHA.108.844506. Epub 2009 May 4. PMID 19414634
- [Background] Ky B, Shults J, Keane MG, Sutton MS, Wolf M, Feldman HI, Reese PP, Anderson CA, Townsend RR, Deo R, Lo J, Gadegbeku C, Carlow D, Sulik MJ, Leonard MB; CRIC Study Investigators. FGF23 modifies the relationship between vitamin D and cardiac remodeling. Circ Heart Fail. 2013 Jul;6(4):817-24. doi: 10.1161/CIRCHEARTFAILURE.112.000105. Epub 2013 Jun 7. PMID 23748358
- [Background] Grabner A, Amaral AP, Schramm K, Singh S, Sloan A, Yanucil C, Li J, Shehadeh LA, Hare JM, David V, Martin A, Fornoni A, Di Marco GS, Kentrup D, Reuter S, Mayer AB, Pavenstadt H, Stypmann J, Kuhn C, Hille S, Frey N, Leifheit-Nestler M, Richter B, Haffner D, Abraham R, Bange J, Sperl B, Ullrich A, Brand M, Wolf M, Faul C. Activation of Cardiac Fibroblast Growth Factor Receptor 4 Causes Left Ventricular Hypertrophy. Cell Metab. 2015 Dec 1;22(6):1020-32. doi: 10.1016/j.cmet.2015.09.002. Epub 2015 Oct 1. PMID 26437603
- [Background] Sabatine MS, Antman EM. The thrombolysis in myocardial infarction risk score in unstable angina/non-ST-segment elevation myocardial infarction. J Am Coll Cardiol. 2003 Feb 19;41(4 Suppl S):89S-95S. doi: 10.1016/s0735-1097(02)03019-x. PMID 12644346
- [Background] O'Connor CM, Hasselblad V, Mehta RH, Tasissa G, Califf RM, Fiuzat M, Rogers JG, Leier CV, Stevenson LW. Triage after hospitalization with advanced heart failure: the ESCAPE (Evaluation Study of Congestive Heart Failure and Pulmonary Artery Catheterization Effectiveness) risk model and discharge score. J Am Coll Cardiol. 2010 Mar 2;55(9):872-8. doi: 10.1016/j.jacc.2009.08.083. PMID 20185037
- [Background] Levy WC, Mozaffarian D, Linker DT, Sutradhar SC, Anker SD, Cropp AB, Anand I, Maggioni A, Burton P, Sullivan MD, Pitt B, Poole-Wilson PA, Mann DL, Packer M. The Seattle Heart Failure Model: prediction of survival in heart failure. Circulation. 2006 Mar 21;113(11):1424-33. doi: 10.1161/CIRCULATIONAHA.105.584102. Epub 2006 Mar 13. PMID 16534009